CLINICAL TRIAL: NCT02860299
Title: Evaluation of Systemic Leakage When a Heparin or Citrate Lock is Injected and Biological and Clinical Repercussions: Ancillary Study of the VERROU-REA Randomized Controlled Trial
Brief Title: Biological and Clinical Measurements Following Systemic Leakage When a Citrate or Heparin Lock is Used
Acronym: VERROU HEMOST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Bovet AOI 2015
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Acute Renal Insufficiency
Keywords: patients
MeSH Terms: conditions — Acute Kidney Injury | interventions — Heparin; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Citrate lock (Experimental)
  Interventions: Drug: citrate 4%; Biological: blood sample
- Heparin lock (Active Comparator)
  Interventions: Drug: unfractionated heparin; Biological: blood sample

INTERVENTIONS:
Drug: citrate 4%
  Arms: Citrate lock
Drug: unfractionated heparin
  Arms: Heparin lock
Biological: blood sample

SUMMARY:
In the VERROUREA study, there were two cases of an abnormal increase in TCA. In theory no leakage of the lock into the bloodstream should have been seen. Lock leakage could have particularly serious, and especially clinical, repercussions in these patients who already have a high risk of haemorrhage given the numerous associated comorbidities. The aim of this study is to investigate the leakage of locks into the bloodstream by measuring, before and after injection of the lock, the evolution of haemostasis tests and calcaemia. The findings will complete safety data already collected in the VERROU REA study.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years
* Requiring dialysis for acute kidney failure
* In whom a first non-tunnelled catheter has been inserted
* In the jugular or femoral position
* Once informed consent has been obtained from the patient, a family member or a person of trust

Exclusion Criteria:

* Patients with active and poorly-controlled bleeding
* Known allergy to citrate
* Liver failure (Factor V <30%)
* Thrombopenia < 30 000/mm3 in the absence of planned corrective measures at the time of randomization
* Known or suspected heparin-induced thrombopenia
* Positive blood cultures without treatment or with inappropriate treatment at the time of randomization
* Catheter inserted in the subclavian position
* Person without national health insurance cover
* Pregnant women
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Level of calcaemia | through study completion an average of 28 days
Level of haemostasis | through study completion an average of 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France